CLINICAL TRIAL: NCT06879041
Title: A Phase I, First-in-human, Dose Escalation Study Of [225Ac]-AZD2284 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Phase I Study of [225Ac]-AZD2284 in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7580C00001
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Dose Escalation Study; Metastatic Prostate Cancer; Radiopharmaceutical; Radiotheranostics; Castration-Resistant Prostate Cancer; Radiotherapy; Six Transmembrane Epithelial Antigen of the Prostate 2 (STEAP2); Actinium; Radioconjugate; Radioligand
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A: Cohort A1: AZD2287 (Hot only) (Experimental): Participants will receive 1 dose of AZD2287. If eligible for treatment, will receive low dose of AZD2284.
  Interventions: Drug: AZD2287; Drug: AZD2284
- Part A: Cohort A2: AZD2275 + AZD2287 (Cold +Hot) (Experimental): Participants will receive low dose of AZD2275 followed by 1 dose of AZD2287. If eligible for treatment, will receive low dose of AZD2284.
  Interventions: Drug: AZD2287; Drug: AZD2275; Drug: AZD2284
- Part A: Cohort A3: AZD2275 + AZD2287 (Cold +Hot) (Experimental): Participants will receive medium dose of AZD2275 followed by 1 dose of AZD2287. If eligible for treatment, will receive low dose of AZD2284.
  Interventions: Drug: AZD2287; Drug: AZD2275; Drug: AZD2284
- Part A Expansion: AZD2287 + AZD2275 (Cold + Hot) (Experimental): Participants will receive dose of AZD2275 determined earlier in the study followed by 1 dose of AZD2287.
  Interventions: Drug: AZD2287; Drug: AZD2275
- Part B (Actinium-225 Dose Escalation): low dose: AZD2284 (Experimental): Participants will receive AZD2287 (± AZD2275 as determined in Part A). If eligible for treatment, will receive low dose of AZD2284.
  Interventions: Drug: AZD2287; Drug: AZD2275; Drug: AZD2284
- Part B (Actinium-225 Dose Escalation): medium dose: AZD2284 (Experimental): Participants will receive AZD2287 (± AZD2275 as determined in Part A). If eligible for treatment, will receive medium dose of AZD2284.
  Interventions: Drug: AZD2287; Drug: AZD2275; Drug: AZD2284
- Part B (Actinium-225 Dose Escalation): high dose 1: AZD2284 (Experimental): Participants will receive AZD2287 (± AZD2275 as determined in Part A). If eligible for treatment, will receive high dose of AZD2284.
  Interventions: Drug: AZD2287; Drug: AZD2275; Drug: AZD2284
- Part B (Actinium-225 Dose Escalation): high dose 2: AZD2284 (Experimental): Participants will receive AZD2287 (± AZD2275 as determined in Part A). If eligible for treatment, will receive high dose of AZD2284.
  Interventions: Drug: AZD2287; Drug: AZD2275; Drug: AZD2284
- Part B: Cohort E1 (Experimental): Participants will receive dose of AZD2284 determined by the earlier results. Expansion cohort may be opened to further characterize the safety and efficacy of the dose level.
  Interventions: Drug: AZD2287; Drug: AZD2275; Drug: AZD2284
- Part B: Cohort E2 (Experimental): Participants will receive dose of AZD2284 determined by the earlier results. Expansion cohort may be opened to further characterize the safety and efficacy of the dose level.
  Interventions: Drug: AZD2287; Drug: AZD2275; Drug: AZD2284

INTERVENTIONS:
Drug: AZD2287 — AZD2287 is administered through intravenous injection.
Drug: AZD2275 — AZD2275 is administered through intravenous infusion.
  Arms: Part A Expansion: AZD2287 + AZD2275 (Cold + Hot); Part A: Cohort A2: AZD2275 + AZD2287 (Cold +Hot); Part A: Cohort A3: AZD2275 + AZD2287 (Cold +Hot); Part B (Actinium-225 Dose Escalation): high dose 1: AZD2284; Part B (Actinium-225 Dose Escalation): high dose 2: AZD2284; Part B (Actinium-225 Dose Escalation): low dose: AZD2284; Part B (Actinium-225 Dose Escalation): medium dose: AZD2284; Part B: Cohort E1; Part B: Cohort E2
Drug: AZD2284 — AZD2284 is administered through intravenous injection.
  Arms: Part A: Cohort A1: AZD2287 (Hot only); Part A: Cohort A2: AZD2275 + AZD2287 (Cold +Hot); Part A: Cohort A3: AZD2275 + AZD2287 (Cold +Hot); Part B (Actinium-225 Dose Escalation): high dose 1: AZD2284; Part B (Actinium-225 Dose Escalation): high dose 2: AZD2284; Part B (Actinium-225 Dose Escalation): low dose: AZD2284; Part B (Actinium-225 Dose Escalation): medium dose: AZD2284; Part B: Cohort E1; Part B: Cohort E2

SUMMARY:
The main purpose of the study is to assess the safety and tolerability of AZD2284, AZD2287, and AZD2275.

DETAILED DESCRIPTION:
This is a first-in-human, Phase I, non-randomized, open-label clinical trial designed to evaluate AZD2284, AZD2287, and AZD2275.

This trial will consist of 2 Parts:

Part A (Imaging):

* Part A (Cold Antibody Exploration): aims to determine the optimal dosing regimen, with or without unconjugated antibody (AZD2275) pre-administration to improve the biodistribution of AZD2287.
* Part A Expansion: aims to explore the prevalence of PSMA and STEAP2 expression by imaging.

Part B (Therapeutic):

* Part B (Actinium-225 Dose Escalation): aims to assess the safety, tolerability, and efficacy of escalating doses of AZD2284 informed by the optimal dosing regimen identified in Part A.
* Part B Expansion Cohorts 1 and 2: aims to explore efficacy of AZD2284.

ELIGIBILITY:
Main Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Histologically confirmed diagnosis of adenocarcinoma of the prostate or neuroendocrine differentiated prostate cancer.
* Must have had prior bilateral orchiectomy and/or ongoing androgen-deprivation therapy and a castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
* At least one metastatic lesion present on baseline Computed Tomography (CT), Magnetic Resonance Imaging (MRI), or bone scan obtained ≤ 28 days prior to the first dose of Investigational Medicinal Product (IMP). Participants may have non-measurable lesions including bone only metastases.
* Adequate organ function

Main Exclusion Criteria:

* Treatment with any radiopharmaceutical within 6 weeks of the first dose of Investigational Medicinal Product (IMP).
* Radiation therapy (RT) within 28 days prior to the first dose and all RT-related events have not recovered to Grade ≤ 1.
* Administration of any systemic cytotoxic or investigational therapy ≤ 28 days of the first dose of IMP or 5 half-lives, whichever is shorter.
* All prior treatment-related adverse events must have resolved to Grade ≤ 1.
* Concurrent severe and/or uncontrolled illness not related to cancer and/or social situation that would limit compliance with study requirements.
* Known or suspected allergies or contraindications to any of the investigational drugs or any component of the investigational drug formulation.
* Clinically relevant proteinuria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 134 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2029-04-16 (Estimated); Study Completion 2029-04-16 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse event (AEs) | Part A: From Screening (Day -28) to Day 28; Part B: Screening (Day -42 to Day -14) up to 5 years
Number of participants with Dose Limiting Toxicities (DLTs) | Part B: Screening (Day -42 to Day -14) up to 2 cycles (84 days) of AZD2284
Estimates of residence time | Part A: Up to Day 8 after dosing with AZD2287 on Day 1
Absorbed radiation doses for AZD2287 and AZD2284 | Part A: Up to Day 8 after dosing with AZD2287 on Day 1; Part B: Up to Day 8 after dosing with AZD2287 on Day -14
Compare organ uptake of AZD2287 with and without pre-dose administration of AZD2275 | Part A: Up to Day 8 after dosing with AZD2287 on Day 1; Part B: Up to Day 8 after dosing with AZD2287 on Day -14
Tumor uptake of AZD2287 in selected regions of interest on SPECT/CT and/or planar images | Part A: Up to Day 8 after dosing with AZD2287 on Day 1; Part B: Up to Day 8 after dosing with AZD2287 on Day -14

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 12 months after the last dose of AZD2284
Proportion of participants with Prostate-Specific Antigen (PSA) 50 | Up to 12 months after the last dose of AZD2284
Proportion of participants with PSA90 | Up to 12 months after the last dose of AZD2284
Time to maximum PSA % decline | Up to 12 months after the last dose of AZD2284
Duration of Response (DoR) | Up to 12 months after the last dose of AZD2284
Radiographic Progression Free Survival (rPFS) | Up to 12 months after the last dose of AZD2284
Overall Survival (OS) | Part A: Up to Day 28; Part B: Up to 5 years
Pharmacokinetic Clearance | Part A: Up to Day 28; Part B: Up to Cycle 2 (each cycle is 42 days)
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Part A: Up to Day 28; Part B: Up to Cycle 2 (each cycle is 42 days)
Maximum observed drug concentration (Cmax) | Part A: Up to Day 28; Part B: Up to Cycle 2 (each cycle is 42 days)
Half-life (t1/2) | Part A: Up to Day 28; Part B: Up to Cycle 2 (each cycle is 42 days)
Changes in plasma concentrations of AZD2287 and AZD2284 following AZD2275 pre-administration compared to AZD2287 and AZD2284 alone | Part A: Up to Day 28; Part B: Up to Cycle 2 (each cycle is 42 days)
Number of participants with positive antidrug antibodies (ADAs) | Part A dose exploration: Up to Day 28; Part B: Up to End of Trial (approximately 1 year)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Omaha, Nebraska
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
- Research Site, East Melbourne, Australia
- South Africa (3):
  - Research Site, CapeTown
  - Research Site, Durban
  - Research Site, Pretoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes",indicatesthat AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/